CLINICAL TRIAL: NCT04891146
Title: The Effect of Inhalation Anesthesia and Total Intravenous Anesthesia on Systemic Inflammatory Immune Index in Major Abdominal Cancer Surgeries
Brief Title: The Effect of Anesthesia on Systemic Inflammatory Immune Index in Major Abdominal Cancer Surgeries
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arsen Güngör, Anesthesiology and Reanimation Specialist, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: AbdurrahmanYAOTRH
Record Dates: First submitted 2021-03-17; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-03

CONDITIONS: Systemic Immune Activation; Cancer Gi; Cancer of Endometrium
MeSH Terms: conditions — Gastrointestinal Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalation anesthesia: Sevoflurane for opioid remifentanyl used
  Interventions: Other: Systemic inflammatory immmune index
- Total Intravenous Anesthesia: Propofol for opioid remifentanyl used
  Interventions: Other: Systemic inflammatory immmune index

INTERVENTIONS:
Other: Systemic inflammatory immmune index — Systemic Inflammatory Immune index calculated from platelet, neutrophil and lymphocyte count

SUMMARY:
The effects of different anesthesia methods on the immune system are variable. In this study, we investigated the effect of inhalation anesthesia and total intravenous anesthesia on the SII value in major abdominal cancer surgeries.

DETAILED DESCRIPTION:
The study was planned prospectively, observationally, on a total of 90 patients who underwent major abdominal cancer surgery. 84 patients were evaluated. The patients were seperated in two groups as inhalation anesthesia and total intravenous anesthesia (TIVA). The demographic data of the patients, type of cancer, type of surgery performed, ASA classification, preoperative chemotherapy intake, preoperative hemogram, postoperative 2nd and 24th hour hemogram, intraoperative and postoperative blood transfusion, and duration of surgery were recorded. Platelet, neutrophil, lymphocyte and SII values were saved.

ELIGIBILITY:
Inclusion Criteria:

* major abdominal cancer surgeries

Exclusion Criteria:

* blood transfusion in last 72 hours
* patients with infection
* hematologic malignancy
* patient controlled analgesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major abdominal cancer patients between 18-85 years included. 40 patients in sevoflurane group and 44 patients in TIVA group collected
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
investigate the effect of anesthesia management on the change of preoperative systemic inflammatory immune index(SII) and postoperative 2.hour and 24.hour SII value | preoperative SII noted, postoperative 2.hour noted and postoperative 24.hour noted
  systemic inflammatory immune index calculated by (platelet x neutrophil)/lymphocyte

CONTACTS AND LOCATIONS:
Overall Officials: Arsen Gungor, Principal Investigator — arsen.gungor@hotmail.com
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Research and Trainee Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
shared after published

REFERENCES:
- [Result] Hu B, Yang XR, Xu Y, Sun YF, Sun C, Guo W, Zhang X, Wang WM, Qiu SJ, Zhou J, Fan J. Systemic immune-inflammation index predicts prognosis of patients after curative resection for hepatocellular carcinoma. Clin Cancer Res. 2014 Dec 1;20(23):6212-22. doi: 10.1158/1078-0432.CCR-14-0442. Epub 2014 Sep 30. PMID 25271081
- [Result] Lee JH, Kang SH, Kim Y, Kim HA, Kim BS. Effects of propofol-based total intravenous anesthesia on recurrence and overall survival in patients after modified radical mastectomy: a retrospective study. Korean J Anesthesiol. 2016 Apr;69(2):126-32. doi: 10.4097/kjae.2016.69.2.126. Epub 2016 Mar 30. PMID 27066202